CLINICAL TRIAL: NCT00448409
Title: A Phase II Trial to Assess the Activity of TroVax® Alone vs. TroVax® Plus Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF) in Patients With Progressive Hormone Refractory Prostate Cancer
Brief Title: Activity of TroVax® Alone vs. TroVax® Plus GM-CSF in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Oxford BioMedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMRI IRB#0106-0009; TV/PHRPC-001/06 (Other: Oxford Biomedica)
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate cancer; hormone refractory prostate cancer; androgen resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — TroVax; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): TroVax alone
  Interventions: Biological: TroVax
- 2 (Experimental): TroVax plus GM-CSF
  Interventions: Biological: TroVax; Drug: GM-CSF

INTERVENTIONS:
Biological: TroVax — 11 Intramuscular injection of TroVax® over 45 weeks. A single dose of 5 x 108 pfu/ml, will be given by an intramuscular injection into the deltoid muscle of the upper arm.
Drug: GM-CSF — 168 subcutaneous GM-CSF injections over 45 weeks. Administered every day as a subcutaneous injection at a dose of 250mcg/m2/d (maximum 500 mcg) in weeks 1 and 2 of each 28 day cycle (total of 14 days per cycle with a total of 12 cycles).
  Other Names: Leukine
  Arms: 2

SUMMARY:
To evaluate the efficacy and safety of Trovax and GM-CSF in patients with prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer is the second leading cause of cancer death in American men. Hormonal ablation, in the form of medical or surgical castration is the cornerstone of management for metastatic prostate cancer however, treatment options for a patient in whom androgen ablation fails are limited. Second-line hormonal agents are generally associated with low response rates and no documented survival benefit.

Historically, chemotherapy was not considered to have significant activity in hormone refractory prostate cancer (HRPCa). This view has changed within the past 10 years, partly because of the availability of prostate-specific antigen (PSA) measurements to monitor tumor burden. Although it seems that chemotherapy, either as a single agent or combination of agents may lead to clinical responses, reduction in PSA measurements, pain control, or improved quality of life, no benefit in overall survival has been definitively proven. The current standard of care for the treatment of metastatic prostate cancer is hormone therapy (androgen blockade).3,4 When this strategy is no longer effective, few good treatment options are left. For this reason, prostate cancer research has aimed to identify new therapeutic modalities to increase the impact of these parameters as well as prolong patient survival.

A total of 24 men with prostate cancer ranging from non-metastatic rising PSA only disease to bony metastatic disease will be enrolled in the study. All patients will have failed androgen treatment and at least one prior taxane chemotherapy or have refused chemotherapy.

Out of the 24 patients, 12 patients will be treated using TroVax® and 12 will be treated using TroVax® plus GM-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* Stable or progressive disease after androgen deprivation.
* Karnofsky Performance Status ≥ 60%.
* At least one prior taxane based chemotherapy for prostate cancer therapy (or patient refusal of chemotherapy)
* At least four weeks have lapsed since prior chemotherapy (if administered)
* Patients on stable doses of bisphosphonates that show subsequent tumor progression may continue on this medication; however, patients are not allowed to initiate bisphosphonate therapy within one month prior to starting therapy or throughout the study.
* Major surgery or radiation therapy completed ≥ 4 weeks prior to enrollment.
* Clinically immunocompetent. All patients are assumed to be immunocompetent unless they have been diagnosed as being immunosuppressed, are receiving oral steroids, immunosuppressive chemotherapy for oncology disorders or are receiving immunosuppressive therapy following transplant.
* Free of clinically apparent autoimmune disease (no prior confirmed diagnosis or treatment for autoimmune disease including Systemic Lupus Erythematosis, Grave's disease, Hashimoto's thyroiditis, multiple sclerosis, insulin dependant diabetes mellitus or systemic (non-joint) manifestations of rheumatoid disease).
* Absolute Lymphocyte Count ≥ 500/µl, ANC >1200/µl, Platelet count >100,000/µl, Hemoglobin > 8 mg/dl
* No evidence of active ischemia on ECG

Exclusion Criteria:

* Patients receiving any other hormonal therapy, including any dose of megestrolacetate (Megace), Proscar (finasteride), any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES), or any systemic corticosteroid must discontinue the agent for at least 4 weeks prior to enrollment. Progressive disease (as defined above) must be documented after discontinuation of the hormonal therapy.
* Patients that initiate bisphosphonate therapy within one month prior to starting therapy or throughout the study.
* No supplements or complementary medicines/botanicals are permitted during the study
* Major surgery or radiation therapy completed ≤ 4 weeks prior to enrollment.
* Prior radiopharmaceuticals (strontium, samarium) within 8 weeks prior to enrollment.
* "Currently active" second malignancy, other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at least less than 30% risk of relapse.
* Serious intercurrent infections or nonmalignant medical illnesses that are uncontrolled.
* Psychiatric illnesses/social situations that would limit compliance with protocol requirements.
* Liver function tests (ALT, AST) more than 1.5 x upper limit of normal (ULN). The bilirubin must be within normal limits.
* Renal function creatinine ≥1.5 x ULN.
* Known allergy to egg proteins.
* Known allergy to neomycin.
* History of allergic response to previous vaccinia vaccinations.
* Chronic oral corticosteroid use (especially anti-emetics) unless prescribed as replacement therapy in the case of adrenal insufficiency.
* Known to test positive for HIV or hepatitis B or C.
* Clinical indication of reduced cardiac function or an ejection fraction of ≤ 40%.
* Requirement for radiotherapy (this is a sign of disease progression and is classed as a withdrawal criterion).
* Concurrent chemotherapy, immunotherapy and radiation therapy
* No investigational or commercial agents or therapies other than those included in protocol treatment may be administered with the intent to treat the patient's malignancy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-05; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
PSA response rate to TroVax® and TroVax® in combination with GM-CSF | restaging every 8 weeks
Anti-5T4 antibody levels | 1st 2 cycles every 2 wks; thereafter about every 4 wks
CD8+ve cellular response to 5T4 antigen as measured by Elispot | at end of study
Assessment of the number of adverse events and serious adverse events in both groups | AEs as occur

SECONDARY OUTCOMES:
Objective response rate | restaging every 8 weeks
Overall survival of the patients | restaging every 8 weeks
Progression-free survival | restaging every 8 weeks
Time to progression | restaging every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No